CLINICAL TRIAL: NCT04512404
Title: Endothelial Microparticles as Potential Biomarkers for Endothelial Dysfunction in Hypercholesterolemia and Its Correlation With Pulse Wave Analysis
Brief Title: Endothelial Microparticles as Potential Biomarkers of Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Nik Nor Izah Nik Ibrahim, Principal Investigator, Universiti Sains Malaysia
Other Study IDs: 1001/PPSP/812211
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- hypercholesterolemia: 3-hydroxy-3-methylglutaric acid coenzyme A (HMG Co-A) reductase inhibitor Types of drug, dosage and frequency is according to the treating physician. This is an observational study.
  Duration of treatment: 3-5 months
  Interventions: Drug: HMG-CoA Reductase Inhibitor

INTERVENTIONS:
Drug: HMG-CoA Reductase Inhibitor
  Other Names: statin

SUMMARY:
Endothelial microparticles (EMP) have a promising role as a diagnostic and prognostic tool in the assessment of endothelial function. This study compares the levels of EMP in hypercholesterolaemia patients before and after treatment with statins and correlates it with the current method of assessing endothelial function using pulse wave analysis.

The current available methods to assess endothelial function are tedious and not suitable to be applied clinically. Detecting EMP levels are simpler as it only involves routine blood taking which is better tolerated by patients.

Outcome from this study will contribute to finding a potential diagnostic, prognostic and treatment assessment tool that is suitable to be used clinically. This will have a large impact in the management of cardiovascular-related disease that is prevalent worldwide and increasing in the developed countries.

DETAILED DESCRIPTION:
General study objective

To evaluate EMP as a simple diagnostic tool in assessing endothelial function in hypercholesterolaemic patients.

Specific objectives:

1. To compare the levels of EMP ( Cluster of differentiation (CD)144, CD62e and CD31+/42-) in hypercholesterolaemics before and after statin.
2. To correlate the levels of EMP with the assessment of endothelial function using pulse wave analysis (PWA) in hypercholesterolaemics before and after statin.

Research design

It is a clinical cohort study involving newly diagnosed hypercholesterolemic patients before and after intervention with statin.

Sampling method and subject recruitment Consecutive sampling of sampling frame will be applied due to limited number of sample who could fulfill the criteria within the planned data collection period.

Data collection method

Screening

Before acceptance into the study, all potential subjects will undergo a screening procedure. A signed written informed consent will be obtained from the subjects before screening procedure is performed. The screening procedure will include detailed history taking on medical history, physical examination and 5 ml venous blood sampling for fasting lipid profile (FLP) from the antecubital vein.

Clinical study session

Once the FLP results are obtained, appointment to attend the clinical study sessions will be arranged with the eligible subjects who fulfil the criteria.

Newly diagnosed hypercholesterolaemia patients recruited will undergo clinical study.

First visit

The first visit will involve blood taking for baseline values, assessment with SphygmoCor and consultation by the treating physician.

During the first visit, 10 ml of venous blood will be withdrawn from the antecubital vein followed by the assessment of endothelial function, augmentation index (AI) and central arterial pressure (CAP) using SphygmoCor.

Venous blood is needed for baseline full blood count (FBC), renal function test (RFT), liver function test (LFT), fasting blood sugar (FBS), high sensitivity C-reactive protein (hs-CRP) and EMP.

Assessment of endothelial function, AI and CAP using SphygmoCor .

Physician consultation

During the first visit, all patients will be seen by the treating physician (a Family Medicine Specialist) at the outpatient clinic (KRK) and advised for therapeutic life style changes (TLC) as recommended by the Malaysian Clinical Practice Guideline (CPG) for Hyperlipidaemia (2011). Patients will be on TLC for a minimum duration of 6 weeks before the next visit.

Second visit

The second visit will only involve blood taking for FLP (5 ml blood) after at least 6 weeks duration of TLC.

Third visit

Once the FLP results are obtained (in approximately a week), patients will then be seen by the treating physician in the clinic.

Patients who do not achieve the targeted LDL level after TLC and indicated for treatment will be prescribed with statin by the attending physician.

Patients who achieve the targeted LDL level after TLC will continue TLC and will be excluded from the study

Fourth visit

The fourth visit will be arranged with the patients 3 months later. 10 ml of blood will be withdrawn for EMP quantification, FLP, hs-CRP and LFT. This will be followed by the assessments of endothelial function, AI and CAP as explained above.

Fourth visit marks the end of the Study 2. Thereafter, patients will continue their treatment at the KRK.

The study duration for each subject will be approximately 5 months.

Patients that miss follow-up or not compliant to the medication prescribed will be excluded from the study analysis. However, this will not compromise the treatment received by patients as they will continue to be treated in KRK.

ELIGIBILITY:
Inclusion Criteria:

1. Hypercholesterolaemia: ( LDL >4.1 mmol/l)
2. Age 35 years and above
3. Agreeable to the treatment with statin if indicated

Exclusion Criteria:

1. Pregnancy and breast feeding
2. Serious medical illness eg kidney failure, liver failure, stroke and malignancy.
3. Arrythmias
4. Contraindicated to statin

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
EMP level and its correlation with endothelial function by pulse wave analysis | 1 day (First visit)
  EMP level: absolute count Endothelial function by pulse wave analysis
EMP level and its correlation with endothelial function by pulse wave analysis | 3 months (Fourth visit)
  EMP level: absolute count Endothelial function by pulse wave analysis

CONTACTS AND LOCATIONS:
Overall Officials: NIk Ibrahim, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia